CLINICAL TRIAL: NCT00121563
Title: Evaluation of TNF-Alpha Modulator for Clinical and Molecular Indicators of Analgesic Effect
Brief Title: Evaluation of a TNF-Alpha Modulator for Clinical and Molecular Indicators of Analgesic Effect
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050193; 05-NR-0193
Record Dates: First submitted 2005-07-20; First posted 2005-07-21 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-02

CONDITIONS: Pain
Keywords: Cytokines; Inflammation; Pain; Injury; Peripheral; Wisdom Teeth; Third Molar Extraction
MeSH Terms: conditions — Pain; Inflammation; Wounds and Injuries | interventions — Thalidomide; Ibuprofen; Diazepam

INTERVENTIONS:
Drug: Thalidomide, Ibuprofen or Diazepam

SUMMARY:
This study will evaluate the role of thalidomide, a tumor necrosis factor (TNF)-alpha modulator, on severe inflammation and relief of pain following extraction of wisdom teeth. TNFs are substances that affect the pathways of pain. This study involves an experimental group in which patients will be given thalidomide or a placebo (an inactive substance); a negative control group receiving the medication diazepam or a placebo; and a positive control group receiving diazepam or ibuprofen.

Patients who are males ages 16 to 35, who are not allergic to aspirin or other nonsteroidal anti-inflammatory drugs (known as NSAIDs), sulfites, or certain anesthetics, and who in good health may be eligible for this study. Females are not eligible, owing to the risks that thalidomide presents to unborn children. To minimize the risk of fetal malformations, male patients who participate must use a condom during sexual intercourse for 4 weeks following the study and must not donate blood for 4 weeks.

The medications used in the study will be given 1 hour before surgery. Then after the wisdom teeth are removed, a small piece of tubing will be placed into both sides of the patient's mouth where the teeth were removed. Every 20 minutes, for the next 6 hours, the researchers will collect inflammatory fluid from the tubing, to measure for changes in anti-inflammatory action. If they request pain relievers, patients will receive the medication ketorolac (Toradol), used for short-term treatment of moderately severe acute pain. Side effects of thalidomide include fatigue, dizziness, and rash. The use of ibuprofen and ketorolac may include the risk of gastrointestinal ulcers and bleeding. Diazepam can cause involuntary muscle movements and drowsiness, as well as dizziness lasting for up to 24 hours after it has been used as sedation. Patients will be instructed not to try to walk alone or to try to drive a vehicle during that period. Other risks related to participation in this study include those usually experienced with removal of wisdom teeth-that is, pain and swelling, bruising from insertion of the sedative into a vein (if needed), possible infection at the extraction site, prolonged bleeding, and numbness.

Benefits from participating are having wisdom teeth removed at no cost as well as close monitoring before and after surgery. Results from the study may help people in the future by improving the management of pain following surgery.

DETAILED DESCRIPTION:
The proposed investigation is a randomized, double-blind, placebo and positive-controlled clinical study to evaluate the role of the cytokine tumor necrosis factor alpha (TNF-alpha) modulator, thalidomide, in acute inflammation and analgesia. The analgesic effect of thalidomide, a putative TNF-alpha modulator, will be evaluated using a model of tissue injury, the oral surgery model. Briefly, healthy males referred for third molar extraction will undergo the surgical extraction of third molars using standard surgical methods. At the completion of the surgical procedure, a microdialysis probe will be placed under the mucogingival flap previously elevated for the surgical procedure and subjects will be observed for pain over the course of six hours following surgery. Thalidomide or control will be administered one hour prior to surgery. Tissue levels of pro-inflammatory cytokines, and inflammatory mediators will be measured at time intervals postoperatively concomitant with pain measurements. Pain will be assessed postoperatively over the course of six hours. Demonstration of amelioration of pain is the primary outcome measure; changes in levels of tissue mediators will be taken as evidence of an acute anti-inflammatory effect of thalidomide. Based on our previous work with the fusion protein etanercept (TNFR:fc) which specifically binds TNF-alpha and prevents its interaction with cellular receptors, similar changes in the inflammatory cascade and clinical endpoints of inflammation may provide insight into the activity of thalidomide on acute inflammation and its clinical sequela, pain.

ELIGIBILITY:
INCLUSION CRITERIA:

* male patients referred for extraction of third molars willing to undergo surgical extraction of all indicated third molars
* a minimum of one partial-bony impacted third molar, with a total difficulty score total of not less than 8
* between the ages of 16 to 35 years (based upon eruption patterns and age-related complications associated with surgical extraction of third molars)
* in good general health- ASA status 1 or 2 (healthy subjects based upon criteria for safe outpatient conscious sedation)
* willing to undergo observation period for six hours postoperatively

EXCLUSION CRITERIA:

* females
* current mental disorder or substance abuse
* allergy to aspirin, NSAIDs, or sulfonamide
* history of peptic ulcers and GI bleeding
* concurrent use of agents which may potentiate the sedative effect of study drugs, alcohol, opioids, benzodiazapines
* chronic use of medications confounding assessment of the inflammatory response or analgesia, antihistamines, NSAIDs, steroids, antidepressants
* presence of chronic debilitating disease (such as diabetes, rheumatoid arthritis, liver disease, etc.)
* presence of symptomatic tooth suggesting infection or inflammation
* excessive surgical difficulty encountered during the surgical procedure, resulting in a difficulty score of 5 for any tooth
* patients with acute narrow angle glaucoma, and open angle glaucoma who are not receiving therapy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2005-07; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Nursing Research (NINR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Anthonsen MW, Solhaug A, Johansen B. Functional coupling between secretory and cytosolic phospholipase A2 modulates tumor necrosis factor-alpha- and interleukin-1beta-induced NF-kappa B activation. J Biol Chem. 2001 Aug 10;276(32):30527-36. doi: 10.1074/jbc.M008481200. Epub 2001 Jun 4. PMID 11390371
- [Background] Barosi G, Grossi A, Comotti B, Musto P, Gamba G, Marchetti M. Safety and efficacy of thalidomide in patients with myelofibrosis with myeloid metaplasia. Br J Haematol. 2001 Jul;114(1):78-83. doi: 10.1046/j.1365-2141.2001.02918.x. PMID 11472348
- [Background] Bastuji-Garin S, Ochonisky S, Bouche P, Gherardi RK, Duguet C, Djerradine Z, Poli F, Revuz J; Thalidomide Neuropathy Study Group. Incidence and risk factors for thalidomide neuropathy: a prospective study of 135 dermatologic patients. J Invest Dermatol. 2002 Nov;119(5):1020-6. doi: 10.1046/j.1523-1747.2002.19502.x. PMID 12445187